CLINICAL TRIAL: NCT05340660
Title: Metabotropic Glutamate Receptor 5 Imaging in Amyotrophic Lateral Sclerosis Using Positron Emission Tomography
Brief Title: mGluR5 Imaging in ALS Using PET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nathalie Braun (Other)
Collaborators: University of Zurich (Other); ETH Zurich (Other)
Responsible Party: Sponsor-Investigator, Nathalie Braun, Principal Investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BASEC Nr. 2021-01044
Record Dates: First submitted 2022-03-29; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Receptor, Metabotropic Glutamate 5; Brain / diagnostic imaging; Positron-Emission Tomography / methods; Radiopharmaceuticals / pharmacokinetics*; PSS232; Humans; Adult
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALS Patient (Experimental)
  Interventions: Radiation: [ 18 F]PSS232

INTERVENTIONS:
Radiation: [ 18 F]PSS232 — [ 18 F]PSS232 for imaging metabotropic glutamate receptor subtype 5 and comparing expression of the receptor in healthy persons and ALS patients

SUMMARY:
In ALS models, it was shown that receptors, that bind an important messenger substance (glutamate) in the brain, are increased. In this research project, the investigators want to use a specific radioactive substance to find out whether these receptors are more detectable in people with ALS than in healthy people and increase over the course of the disease.

DETAILED DESCRIPTION:
With this study, the investigators want to examine whether receptors (docking points on the surface of a nerve cell) that bind an important messenger substance in the brain (glutamate) are increased in patients with amyotrophic lateral sclerosis (ALS) as the disease progresses. Based on observations from ALS models, the investigators suspect that this increase in receptors contributes to the damage to the nerve cells in ALS.

To image these receptors, the investigators use a specific radioactive substance and imaging combining positron emission tomography (PET), magnetic resonance spectroscopy (MRS) and magnetic resonance imaging (MRI) of the brain and spinal cord.

The investigators will examine healthy people and ALS patients. The reason is that little is known about the receptor, even in healthy people. The investigators also do not know if and when the receptor is increasingly detectable in the course of the ALS disease. Only by comparing diseased and healthy people it can be determined if and when the receptor is built up in ALS patients. The investigators also hope to gain more information, e.g. about the distribution of receptors in the brain of healthy people compared to patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically probable, probable laboratory supported, or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria (EEC) (45)
* Disease duration ≤18 months
* Pre-study ALSFRS-R progression between disease onset and screening of - 0.4 points/month or worse (calculated by ALSFRS -R total score decline form 48 divided by the months since onset of ALS symptoms)
* Upright slow vital capacity (sVC) ≥65 % of normal (best of three measurements)

Exclusion Criteria :

* Previous participation in another clinical study involving trial medication within the preceding 12 weeks
* History or presence of significant psychiatric disease, such as depression, evaluated with the ALS depression questionnaire (ADI-12) ≥ 23 (43) since depression has an impact on mGluR5 expression (44)
* Use of tobacco, including cigarettes, smokeless tobacco, cigars, and pipes; Ex- smoker having quit smoking ≥ 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in [18F]PSS232 uptake in the brain and spinal cord in ALS patients at 6 months | Baseline and 6 months
  Difference of [18F]PSS232 uptake in the brain and spinal cord of ALS patients at baseline and day 180, as assessed by PET and MRI to allow morphological mapping.

SECONDARY OUTCOMES:
Difference of [18F]PSS232 uptake in the brain and spinal cord between ALS patients and healthy, age and gender-matched subjects. | 6 months
  Difference of [18F]PSS232 uptake in the brain and spinal cord of ALS patients and healthy subjects at baseline and day 180, as assessed by PET and MRI to allow morphological mapping
Correlation of change from baseline of [18F]PSS232 uptake with change from baseline of ALSFRS-R Score at day 180 | 6 months
  Change from baseline to day 180 in [18F]PSS232 uptake in the brain and spinal cord in ALS patients will be correlated to change from baseline to 180d in the ALS Functional Rating Scale (ALSFRS-R), evaluating bulbar, respiratory, upper limb and lower limb function with a total score of 48 (minimal value 0, maximal value 48, higher scores mean a better outcome).
Correlation of change from baseline of [18F]PSS232 uptake with change from baseline of respiratory function, as measuerd by slow vital capacity (sVC) and sniff nasal inspiratory pressure (SNIP) at day 180 | 6 months
  Change from baseline to day 180 in [18F]PSS232 uptake in the brain and spinal cord in ALS patients will be correlated to change from baseline to 180d in respiratory function, as measured by slow vital capacity (sVC) and sniff nasal inspiratory pressure (SNIP).
Correlation of change from baseline of [18F]PSS232 uptake with change from baseline of ECAS at day 180 | 6 months
  Change from baseline to day 180 in [18F]PSS232 uptake in the brain and spinal cord in ALS patients will be correlated to change from baseline to 180d in cognitive and behavioral function, as assessed by Edinburgh cognitive and behavioral ALS Screen (ECAS, minimal value 0, maximal value 136, higher scores mean a better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Braun, MD, PhD, Principal Investigator — Neuromuscular Center/ALS Clinic, Cantonal Hospital St. Gallen, 9007 St. Gallen, Switzerland
Locations (1):
- Neuromuscular Center/ALS Clinic, Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland